CLINICAL TRIAL: NCT02952820
Title: A Long-Term Multicenter, Randomized, Double-Blind, Controlled, Parallel Group Study of the Safety and Efficacy of Lemborexant in Subjects With Insomnia Disorder (SUNRISE 2)
Brief Title: Long-term Study of Lemborexant in Insomnia Disorder (SUNRISE 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2006-G000-303; 2015-001463-39 (EudraCT Number)
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2017-12

CONDITIONS: Insomnia Disorder
Keywords: insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — lemborexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (3):
- lemborexant 5 milligrams (mg) (Experimental): Lemborexant 5 mg will be taken orally in tablet form at home each night immediately before the time the participant intends to try to sleep.
  Interventions: Drug: lemborexant
- lemborexant 10 mg (Experimental): Lemborexant 10 mg will be taken orally in tablet form at home each night immediately before the time the participant intends to try to sleep.
  Interventions: Drug: lemborexant
- Placebo matched to lemborexant (Placebo Comparator): Lemborexant-matched placebo will be taken orally in tablet form at home each night immediately before the time the participant intends to try to sleep.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lemborexant
  Arms: lemborexant 10 mg; lemborexant 5 milligrams (mg)
Drug: Placebo
  Arms: Placebo matched to lemborexant

SUMMARY:
The key objectives of this study are to determine, using sleep diaries, whether lemborexant at the doses 5 milligrams (mg) and 10 mg is superior to placebo on subjective sleep onset, subjective sleep efficiency, and subjective sleep maintenance in participants with insomnia disorder.

DETAILED DESCRIPTION:
This is a long-term (approximately 1 year), multicenter, randomized, controlled, double-blind, parallel group study of two doses of lemborexant and placebo in approximately 900 male or female participants with insomnia disorder. Approximately 40% of participants will be age 65 years or older. The study will last a maximum of 60 weeks, and will include a Screening Period, an approximately 54-week Treatment Period (during which study medication will be administered), and a 2-week Follow-up Period. All participants will receive lemborexant for at least 6 months and will receive placebo at some point during the study. Participants will not know which medication they receive (lemborexant or placebo) until the study has been completed, and will not know the timings at which the medication will change.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older at the time of informed consent
* Meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM 5) criteria for Insomnia Disorder, as follows:

  * Complains of dissatisfaction with nighttime sleep in the form of difficulty getting to sleep, difficulty staying asleep, and/or awakening earlier in the morning than desired despite adequate opportunity for sleep
  * Frequency of complaint ≥3 times per week
  * Duration of complaint ≥3 months
  * Associated with complaint of daytime impairment
* History of (Subjective Sleep Onset Latency) sSOL ≥30 minutes on at least 3 nights per week in the previous 4 weeks and/or subjective Wake after Sleep Onset (sWASO) ≥60 minutes on at least 3 nights per week in the previous 4 weeks
* History of regular time spent in bed, either sleeping or trying to sleep, between 7 and 9 hours
* Regular bedtime, between 21:00 and 01:00 and regular wake time, the time the participant gets out of bed for the day, between 05:00 and 10:00
* Insomnia Severity Index (ISI) score ≥15
* Confirmation of current insomnia symptoms as determined from the Sleep Diary completed on at least 7 consecutive mornings (minimum 5 of 7 for eligibility), such that sSOL ≥30 minutes on at least 3 of the 7 nights and/or sWASO ≥60 minutes on at least 3 of the 7 nights
* Confirmation of time spent in bed, as determined from on the Sleep Diary completed on 7 mornings between the first and second screening visit, such that there are not more than 2 nights with duration of time spent in bed 7 hours and 10 hours
* Confirmation of regular bedtimes and wake times such that the participant has a regular time spent in bed, either sleeping or trying to sleep, between 7 and 10 hours for the final 7 nights of the before visit 3.
* Confirmation of regular bedtime between 21:00 and 01:00 and time of getting out of bed for the day between 05:00 and 10:00 for the final 7 nights of the before visit 3.
* Willing and able to comply with all aspects of the protocol, including staying in bed for at least 7 hours each night
* Willing to not start a behavioral or other treatment program for insomnia during the participants participation in the study

Exclusion Criteria:

* A current diagnosis of sleep-related breathing disorder, periodic limb movement disorder, restless legs syndrome, circadian rhythm sleep disorder, or an exclusionary score on screening instruments to rule out individuals with symptoms of certain sleep disorders other than insomnia.

  * STOPBang score greater than or equal to (>=) 5
  * International Restless Legs Scale (IRLS) score >=16
  * Epworth Sleepiness Scale (ESS) score >15
* Reports symptoms potentially related to narcolepsy that in the clinical opinion of the investigator indicates the need for referral for a diagnostic evaluation for the presence of narcolepsy
* Reports a history of sleep-related violent behavior, or sleep driving, or any other complex sleep-related behavior, eg, making phone calls, or preparing and eating food while asleep
* For participants who underwent polysomnography (PSG) within the previous year:

  * Age 18 to 64 years: Apnea Hypopnea Index ≥10, or Periodic Limb Movements with Arousal Index ≥10
  * Age ≥65 years: Apnea Hypopnea Index >15, or Periodic Limb Movements with Arousal Index >15
* Beck Depression Inventory - II (BDI II) score >19 at Screening
* Beck Anxiety Inventory (BAI) score >15 at Screening
* Habitually naps more than 3 times per week
* Females who are breastfeeding or pregnant at Screening or Study Baseline
* Females of childbearing potential who are not practicing acceptable pregnancy prevention methods (NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal or have been sterilized surgically.)
* Excessive caffeine use that in the opinion of the investigator contributes to the participant's insomnia, or habitually consumes caffeine-containing beverages after 18:00 and is unwilling to forego caffeine after 18:00 for the duration of his/her participation in the study
* History of drug or alcohol dependency or abuse within approximately the previous 2 years
* Reports habitually consuming more than 14 drinks containing alcohol per week (females) or more than 21 drinks containing alcohol per week (males), or unwilling to limit alcohol intake to no more than 2 drinks per day or forego having alcohol within the 3 hours before bedtime for the duration of his/her participation in the study
* A prolonged QT/QT interval corrected by Fridericia's formula (QTcF >450 ms) as demonstrated by a repeated electro cardiogram(ECG) at Screening (repeated only if initial ECG indicates a QTcF interval >450 ms)
* Current evidence of clinically significant disease (e.g., cardiac, respiratory, gastrointestinal, renal, neurological [including participants who lack capacity and/or whose cognitive decline indicates disorientation to person/place/time and/or situation], or psychiatric disease or malignancy other than basal cell carcinoma) or chronic pain that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments
* Comorbid nocturia resulting in frequent need to get out of bed to use the bathroom during the night
* Scheduled for major surgery during the study
* Used any prohibited prescription or over-the-counter concomitant medications within 1 week before the first dose of study medication
* Used any modality of treatment for insomnia, including cognitive behavioral therapy or marijuana within 2 weeks before Screening
* Failed treatment with suvorexant (Belsomra®) (efficacy and/or safety) following treatment with an appropriate dose and of adequate duration in the opinion of the investigator
* Transmeridian travel across more than 3 time zones in the 2 weeks before Screening, or between Screening and Study Baseline
* Previously participated in any clinical trial of lemborexant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 971 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eisai Medical Information, Study Director — Eisai Inc.
Locations (114):
- United States (42):
  - Facility # 1, Chandler, Arizona
  - Facility # 2, Chandler, Arizona
  - Facility # 1, Rogers, Arkansas
  - Facility # 1, Beverly Hills, California
  - Facility # 2, Los Angeles, California
  - Facility # 1, Los Angeles, California
  - Facility # 1, Redlands, California
  - Facility # 1, Sacramento, California
  - Facility # 1, Santa Monica, California
  - Facility # 1, Torrance, California
  - Facility # 1, Colorado Springs, Colorado
  - Facility # 1, Celebration, Florida
  - Facility # 1, Hialeah, Florida
  - Facility # 1, Homestead, Florida
  - Facility # 1, Jacksonville, Florida
  - Facility # 1, Lauderhill, Florida
  - Facility # 1, Maitland, Florida
  - Innovative Clinical Research Inc, Miami, Florida
  - Facility # 1, Ocala, Florida
  - Facility # 1, Orlando, Florida
  - Facility # 1, Oviedo, Florida
  - Facility # 1, Pinellas Park, Florida
  - Facility # 1, Tampa, Florida
  - Facility # 1, The Villages, Florida
  - Facility # 1, Evansville, Indiana
  - Facility # 1, Elkridge, Maryland
  - Facility # 1, Quincy, Massachusetts
  - Facility # 1, Kansas City, Missouri
  - Facility # 1, Albuquerque, New Mexico
  - Facility # 1, Brooklyn, New York
  - Facility # 1, Hickory, North Carolina
  - Facility # 1, Dayton, Ohio
  - Facility # 2, Oklahoma City, Oklahoma
  - Facility # 1, Oklahoma City, Oklahoma
  - Facility # 1, Portland, Oregon
  - Facility # 1, Lincoln, Rhode Island
  - Facility # 1, Memphis, Tennessee
  - Facility # 1, Austin, Texas
  - Facility # 2, Austin, Texas
  - Facility # 1, Fort Worth, Texas
  - Facility # 1, San Angelo, Texas
  - Facility # 1, Seattle, Washington
- Canada (4):
  - Facility # 1, Kelowna, British Columbia
  - Facility # 1, Toronto, Ontario
  - Facility # 1, Point-Claire, Quebec
  - Facility # 1, Sherbrooke, Quebec
- Finland (6):
  - Facility # 1, Oulu, Oulun Laani
  - Facility # 1, Helsinki
  - Facility # 1, Kuopio
  - Facility # 1, Tampere
  - Facility # 1, Turku
  - Facility # 2, Turku
- Germany (7):
  - Facility # 1, Bochum, North Rhine-Westphalia
  - Facility # 1, Leipzig, Saxony
  - Facility # 1, Berlin
  - Facility # 2, Berlin
  - Facility # 3, Berlin
  - Facility # 1, Hamburg
  - Facility # 1, Hanover
- Italy (3):
  - Facility # 1, Milan, Lombardy
  - Facility # 1, Siena, Tuscany
  - Facility # 1, Roma
- Japan (24):
  - Eisai Trail Site 1, Maebashi, Gunma
  - Eisai Trail Site 1, Sapporo, Hokkaido
  - Eisai Trail Site 2, Sapporo, Hokkaido
  - Eisai Trail Site 3, Sapporo, Hokkaido
  - Eisai Trail Site 4, Sapporo, Hokkaido
  - Eisai Trail Site 1, Sagamihara, Kanagawa
  - Eisai Trial Site 1, Yokohama, Kanagawa
  - Eisai Trial Site 2, Yokohama, Kanagawa
  - Eisai Trial Site 3, Yokohama, Kanagawa
  - Eisai Trail Site 1, Tokorozawa, Saitama
  - Eisai Trail Site 1, Arakawa City, Tokyo
  - Eisai Trail Site 1, Katsushika-ku, Tokyo
  - Eisai Trail Site 1, Minato, Tokyo
  - Eisai Trail Site 2, Minato, Tokyo
  - Eisai Trail Site 1, Musashino, Tokyo
  - Eisai Trail Site 1, Ōta-ku, Tokyo
  - Eisai Trail Site 2, Ōta-ku, Tokyo
  - Eisai Trail Site 3, Ōta-ku, Tokyo
  - Eisai Trail Site 1, Shibuya City, Tokyo
  - Eisai Trail Site 1, Shinagawa, Tokyo
  - Eisai Trail Site 2, Shinagawa, Tokyo
  - Eisai Trail Site 1, Shinjuku, Tokyo
  - Eisai Trail Site 2, Shinjuku, Tokyo
  - Eisai Trail Site 1, Toshima City, Tokyo
- Facility # 1, Monterrey, Nuevo León, Mexico
- New Zealand (5):
  - Facility # 1, Wellington, North Island
  - Facility # 1, Christchurch, South Island
  - Facility # 1, Dunedin, South Island
  - Facility # 1, Auckland
  - Facility # 1, Rotorua
- Poland (7):
  - Facility # 1, Tarnów, Lesser Poland Voivodeship
  - Facility # 1, Warsaw, Masovian Voivodeship
  - Facility # 1, Gdansk
  - Facility # 1, Katowice
  - Facility # 1, Ostróda
  - Facility # 2, Warsaw
  - Facility # 3, Warsaw
- Romania (5):
  - Facility # 1, Brasov
  - Facility # 1, Bucharest
  - Facility # 1, Constanța
  - Facility # 1, Sibiu
  - Facility # 1, Târgu Mureş
- South Korea (5):
  - Facility # 1, Seongnam-si, Gyeonggido
  - Facility # 1, Suwon, Gyeonggido
  - Facility # 1, Daegu
  - Facility # 1, Seoul
  - Facility # 3, Seoul
- Spain (5):
  - Facility # 1, Palma de Mallorca, Balearic Islands
  - Facility # 1, Torrejón de Ardoz, Madrid
  - Facility # 1, Quart de Poblet, Valencia
  - Facility # 1, Barcelona
  - Facility # 1, Valencia

REFERENCES:
- [Derived] Chepke C, Cote KA, Pinner K, Yardley J, Lundwall C, Moline M. Effect of Lemborexant on Daytime Functioning in Adults With Insomnia: Patient-Reported Outcomes From a Phase 3 Clinical Trial. Prim Care Companion CNS Disord. 2025 Jan 16;27(1):24m03810. doi: 10.4088/PCC.24m03810. PMID 39823487
- [Derived] Arnold V, Ancoli-Israel S, Dang-Vu TT, Mishima K, Pinner K, Malhotra M, Moline M. Efficacy of Lemborexant in Adults >/= 65 Years of Age with Insomnia Disorder. Neurol Ther. 2024 Aug;13(4):1081-1098. doi: 10.1007/s40120-024-00622-9. Epub 2024 May 15. PMID 38748321
- [Derived] Citrome L, Juday TR, Lundwall C. Lemborexant and Daridorexant for the Treatment of Insomnia: An Indirect Comparison Using Number Needed to Treat, Number Needed to Harm, and Likelihood to Be Helped or Harmed. J Clin Psychiatry. 2023 Oct 2;84(6):23m14851. doi: 10.4088/JCP.23m14851. PMID 37796657
- [Derived] Terauchi M, Cheng JY, Yardley J, Pinner K, Moline M, Malhotra M, Inabe K, Nishida M, Pappadopulos E. Efficacy and safety of lemborexant in midlife women with insomnia disorder. Menopause. 2023 Aug 1;30(8):839-848. doi: 10.1097/GME.0000000000002209. Epub 2023 Jun 20. PMID 37339396
- [Derived] Dash A, Pinner K, Inoue Y, Hayashida K, Lim SC, Yun CH, Lan TH, Huang CL, Yardley J, Kubota N, Moline M. Efficacy and safety of lemborexant over 12 months in Asian adults with insomnia disorder. Sleep Med X. 2022 Mar 24;4:100044. doi: 10.1016/j.sleepx.2022.100044. eCollection 2022 Dec. PMID 35402894
- [Derived] Chepke C, Jain R, Rosenberg R, Moline M, Yardley J, Pinner K, Kumar D, Perdomo C, Filippov G, Atkins N, Malhotra M. Improvement in fatigue and sleep measures with the dual orexin receptor antagonist lemborexant in adults with insomnia disorder. Postgrad Med. 2022 Apr;134(3):316-325. doi: 10.1080/00325481.2022.2049553. Epub 2022 Mar 20. PMID 35254948
- [Derived] Roth T, Rosenberg R, Morin CM, Yardley J, Pinner K, Perdomo C, Atkins N Jr, Pappadopulos E, Malhotra M, Moline M. Impact of lemborexant treatment on insomnia severity: analyses from a 12-month study of adults with insomnia disorder. Sleep Med. 2022 Feb;90:249-257. doi: 10.1016/j.sleep.2022.01.024. Epub 2022 Feb 8. PMID 35220140
- [Derived] Citrome L, Juday T, Frech F, Atkins N Jr. Lemborexant for the Treatment of Insomnia: Direct and Indirect Comparisons With Other Hypnotics Using Number Needed to Treat, Number Needed to Harm, and Likelihood to Be Helped or Harmed. J Clin Psychiatry. 2021 Jun 1;82:20m13795. doi: 10.4088/JCP.20m13795. PMID 34077032
- [Derived] Yardley J, Karppa M, Inoue Y, Pinner K, Perdomo C, Ishikawa K, Filippov G, Kubota N, Moline M. Long-term effectiveness and safety of lemborexant in adults with insomnia disorder: results from a phase 3 randomized clinical trial. Sleep Med. 2021 Apr;80:333-342. doi: 10.1016/j.sleep.2021.01.048. Epub 2021 Feb 1. PMID 33636648
- [Derived] Inoue Y, Watanabe T, Takashima S, Takase T, Ishikawa K, Kubota N, Yardley J, Moline M. Efficacy and safety of lemborexant in adults with insomnia: comparing Japanese and non-Japanese subgroups from the global, phase 3, randomized, double-blind, placebo-controlled SUNRISE 2 study. J Clin Sleep Med. 2021 May 1;17(5):1067-1074. doi: 10.5664/jcsm.9148. PMID 33576735
- [Derived] Karppa M, Yardley J, Pinner K, Filippov G, Zammit G, Moline M, Perdomo C, Inoue Y, Ishikawa K, Kubota N. Long-term efficacy and tolerability of lemborexant compared with placebo in adults with insomnia disorder: results from the phase 3 randomized clinical trial SUNRISE 2. Sleep. 2020 Sep 14;43(9):zsaa123. doi: 10.1093/sleep/zsaa123. PMID 32585700

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 119 investigative sites in Japan, Korea, Finland, Germany, Italy, New Zealand, Poland, Romania, Spain, Canada, Mexico, and the United States from 15 November 2016 to 08 January 2019.
Pre-assignment Details: A total of 2059 participants were screened, of which 1088 were screen failures and 971 participants were randomized to receive study treatment.
Groups:
- Placebo: Participants received lemborexant-matched placebo, tablet, orally, once daily for up to Month 6 in the placebo-controlled treatment period. Then they were re-randomized to lemborexant 5 milligram (mg) or lemborexant 10 mg up to Month 12.
- Lemborexant 5 mg: Participants received lemborexant 5 mg, tablets, orally, once daily through Month 1-6 (in Period 1) and Month 7-12 (in Period 2).
- Lemborexant 10 mg: Participants received lemborexant 10 mg, tablets, orally, once daily through Month 1-6 (in Period 1) and Month 7-12 (in Period 2).
Period: Placebo-Controlled Treatment (6 Months)
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Started | 325 | 323 | 323
Treated | 321 | 319 | 319
Safety Analysis Set | 319 | 314 | 314
Completed | 261 | 254 | 235
Not Completed | 64 | 69 | 88
Not completed — Adverse Event | 8 | 9 | 16
Not completed — Lost to Follow-up | 7 | 7 | 6
Not completed — Subject choice | 15 | 12 | 17
Not completed — Inadequate therapeutic effect | 17 | 12 | 11
Not completed — Other than specified | 0 | 14 | 13
Not completed — Withdrawal of consent | 13 | 11 | 21
Not completed — Not treated | 4 | 4 | 4
Period: Active Treatment Period (6 Months)
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Started | 0 (Participants from Placebo were re-randomized to Lemborexant 5 mg and Lemborexant 10 mg.) | 384 | 352
Completed | 0 | 346 | 321
Not Completed | 0 | 38 | 31
Not completed — Adverse Event | 0 | 6 | 5
Not completed — Lost to Follow-up | 0 | 4 | 6
Not completed — Subject choice | 0 | 10 | 7
Not completed — Inadequate therapeutic effect | 0 | 6 | 2
Not completed — Withdrawal of consent | 0 | 6 | 8
Not completed — Other than specified | 0 | 6 | 2
Not completed — Not treated | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) was the group of randomized participants who received at least 1 dose of randomized study drug and had at least 1 postdose primary efficacy measurement.
Groups:
- Placebo: Participants received lemborexant-matched placebo, tablet, orally, once daily for up to Month 6 in the placebo-controlled treatment period. Then they were re-randomized to lemborexant 5 mg or lemborexant 10 mg up to Month 12.
- Total: Total of all reporting groups
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg | Total
Number analyzed (Participants) | 318 | 316 | 315 | 949
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (14.01) | 54.2 (13.74) | 54.8 (13.68) | 54.5 (13.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 209 | 222 | 647
  Male | 102 | 107 | 93 | 302
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 19 | 19 | 72
  Not Hispanic or Latino | 284 | 297 | 296 | 877
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 232 | 222 | 225 | 679
  Black or African American | 23 | 27 | 26 | 76
  Japanese | 54 | 53 | 54 | 161
  Chinese | 0 | 3 | 1 | 4
  Other Asian | 5 | 5 | 3 | 13
  American Indian or Alaska Native | 0 | 1 | 2 | 3
  Native Hawaiian or other Pacific Islander | 0 | 1 | 0 | 1
  Other | 4 | 4 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Subjective Sleep Onset Latency (sSOL) at Month 6
Description: sSOL was defined as estimated minutes from the time that the participant attempted to sleep until sleep onset.
Time Frame: Baseline and Month 6
Population: The FAS was the group of randomized participants who received at least one dose of randomized study drug and had at least one postdose primary efficacy measurement. Number analyzed refers to participants evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 318 | 316 | 315
minutes
  Baseline: number analyzed (Participants) | 316 | 314 | 312
  Baseline | 64.03 (45.209) | 62.19 (45.674) | 64.97 (44.020)
  Change at Month 6: number analyzed (Participants) | 249 | 245 | 229
  Change at Month 6 | -16.57 (35.313) | -29.39 (33.261) | -32.49 (35.962)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; Analysis was based on mixed effect model repeated measurement analysis (MMRM) model with log transformation of sSOL and factors for age group, region, treatment, visit (Month 6), and treatment-by-visit interaction as fixed effects, and the study baseline sSOL as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (missing not at random/complete case missing value [MNAR/CCMV]); Test type: Superiority; p < .0001, Mixed Models Analysis; least squares geometric mean (LSGM)ratio = 0.732, 95% CI 2-sided [0.636 to 0.843]
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; Analysis was based on MMRM model with log transformation of sSOL and factors for age group, region, treatment, visit (Month 6), and treatment-by-visit interaction as fixed effects, and the study baseline sSOL as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p < .0001, Mixed Models Analysis; LSGM ratio = 0.701, 95% CI 2-sided [0.607 to 0.810]

2. Secondary Outcome: Change From Baseline in sSOL at the Beginning of Treatment (Mean of the 7 Nights After the First Dose in Placebo-Controlled Period), and at Months 1 and 3
Description: sSOL was defined as estimated minutes from time attempted to sleep to sleep onset.
Time Frame: Baseline, (mean of 7 nights [approximately Week 1]), Months 1 and 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 318 | 316 | 315
minutes
  Baseline: number analyzed (Participants) | 316 | 314 | 312
  Baseline | 64.03 (45.209) | 62.19 (45.674) | 64.97 (44.020)
  Change at 1st 7 nights: number analyzed (Participants) | 314 | 310 | 310
  Change at 1st 7 nights | -4.11 (27.671) | -16.86 (27.784) | -18.89 (31.003)
  Change at Month 1: number analyzed (Participants) | 299 | 298 | 297
  Change at Month 1 | -11.48 (32.726) | -19.41 (32.221) | -24.06 (35.234)
  Change at Month 3: number analyzed (Participants) | 279 | 268 | 264
  Change at Month 3 | -13.84 (35.277) | -25.08 (34.081) | -27.94 (39.192)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; First 7 nights after the first dose (Statistical analysis 1): Based on MMRM model with log transformation of sSOL and factors for age group, region, treatment, visit (First 7 nights), and treatment-by-visit interaction as fixed effects, and the study baseline sSOL as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p < .0001, Mixed Models Analysis; LSGM ratio = 0.781, 95% CI 2-sided [0.725 to 0.842]
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; First 7 nights after the first dose (Statistical analysis 2): Based on MMRM model with log transformation of sSOL and factors for age group, region, treatment, visit (First 7 nights), and treatment-by-visit interaction as fixed effects, and the study baseline sSOL as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p < .0001, Mixed Models Analysis; LSGM ratio = 0.752, 95% CI 2-sided [0.698 to 0.811]
Statistical Analysis 3: Comparison: Placebo vs Lemborexant 5 mg; Month 1 (Statistical analysis 3): Based on MMRM model with log transformation of sSOL and factors for age group, region, treatment, visit (Month 1), and treatment-by-visit interaction as fixed effects, and the study baseline sSOL as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p < .0001, Mixed Models Analysis; LSGM ratio = 0.810, 95% CI 2-sided [0.735 to 0.893]
Statistical Analysis 4: Comparison: Placebo vs Lemborexant 10 mg; Month 1 (Statistical analysis 4): Based on MMRM model with log transformation of sSOL and factors for age group, region, treatment, visit (Month 1), and treatment-by-visit interaction as fixed effects, and the study baseline sSOL as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p < .0001, Mixed Models Analysis; LSGM ratio = 0.770, 95% CI 2-sided [0.698 to 0.848]
Statistical Analysis 5: Comparison: Placebo vs Lemborexant 5 mg; Month 3 (Statistical analysis 5): Based on MMRM model with log transformation of sSOL and factors for age group, region, treatment, visit (Month 3), and treatment-by-visit interaction as fixed effects, and the study baseline sSOL as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p < .0001, Mixed Models Analysis; LSGM ratio = 0.778, 95% CI 2-sided [0.690 to 0.878]
Statistical Analysis 6: Comparison: Placebo vs Lemborexant 10 mg; Month 3 (Statistical analysis 6): Based on MMRM model with log transformation of sSOL and factors for age group, region, treatment, visit (Month 3), and treatment-by-visit interaction as fixed effects, and the study baseline sSOL as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p < .0001, Mixed Models Analysis; LSGM ratio = 0.770, 95% CI 2-sided [0.681 to 0.869]

3. Secondary Outcome: Change From Baseline in Subjective Sleep Efficiency (sSE) at the Beginning of Treatment (Mean of the 7 Nights After the First Dose in Placebo-Controlled Period), and at Months 1, 3 and 6
Description: sSE was defined as percentage of subjective total sleep time (sTST) divided by subjective time spent in bed, calculated as the interval from the time the participant reported attempting to sleep until the time participant stopped trying to sleep for the night (operationalized as the time the participant got out of bed for the day), and time spent asleep derived from subjective time spent in bed minus sWASO.
Time Frame: Baseline, (mean of 7 nights [approximately Week 1]), Months 1, 3 and 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of sTST
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 318 | 316 | 315
percentage of sTST
  Baseline: number analyzed (Participants) | 307 | 302 | 299
  Baseline | 61.34 (17.836) | 63.14 (18.231) | 62.03 (17.248)
  Change at 1st 7 nights: number analyzed (Participants) | 303 | 295 | 296
  Change at 1st 7 nights | 2.68 (10.765) | 6.61 (10.386) | 8.27 (10.566)
  Change at Month 1: number analyzed (Participants) | 291 | 284 | 282
  Change at Month 1 | 6.11 (12.876) | 7.87 (12.263) | 9.92 (12.922)
  Change at Month 3: number analyzed (Participants) | 269 | 256 | 251
  Change at Month 3 | 9.16 (13.644) | 13.03 (13.522) | 13.61 (14.035)
  Change at Month 6: number analyzed (Participants) | 242 | 235 | 220
  Change at Month 6 | 10.36 (13.799) | 15.34 (14.613) | 15.55 (15.617)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; First 7 nights (Statistical analysis 1): Based on MMRM model with factors of age group, region, treatment, visit (First 7 nights), and treatment-by-visit interaction as fixed effect, and the study baseline sSE as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p < .0001, Mixed Models Analysis; LSM Difference = 4.299, 95% CI 2-sided [2.638 to 5.961], Standard Error of Mean 0.848
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; First 7 nights (Statistical analysis 2): Based on MMRM model with factors of age group, region, treatment, visit (First 7 nights), and treatment-by-visit interaction as fixed effect, and the study baseline sSE as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p < .0001, Mixed Models Analysis; LSM Difference = 5.793, 95% CI 2-sided [4.133 to 7.452], Standard Error of Mean 0.846
Statistical Analysis 3: Comparison: Placebo vs Lemborexant 5 mg; Month 1 (Statistical analysis 3): Based on MMRM model with factors of age group, region, treatment, visit (Month 1), and treatment-by-visit interaction as fixed effect, and the study baseline sSE as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p = 0.0230, Mixed Models Analysis; LSM Difference = 2.227, 95% CI 2-sided [0.307 to 4.146], Standard Error of Mean 0.979
Statistical Analysis 4: Comparison: Placebo vs Lemborexant 10 mg; Month 1 (Statistical analysis 4): Based on MMRM model with factors of age group, region, treatment, visit (Month 1), and treatment-by-visit interaction as fixed effect, and the study baseline sSE as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p = 0.0003, Mixed Models Analysis; LSM Difference = 3.615, 95% CI 2-sided [1.635 to 5.595], Standard Error of Mean 1.010
Statistical Analysis 5: Comparison: Placebo vs Lemborexant 5 mg; Month 3 (Statistical analysis 5): Based on MMRM model with factors of age group, region, treatment, visit (Month 3), and treatment-by-visit interaction as fixed effect, and the study baseline sSE as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p = 0.0001, Mixed Models Analysis; LSM Difference = 4.222, 95% CI 2-sided [2.068 to 6.377], Standard Error of Mean 1.099
Statistical Analysis 6: Comparison: Placebo vs Lemborexant 10 mg; Month 3 (Statistical analysis 6): Based on MMRM model with factors of age group, region, treatment, visit (Month 3), and treatment-by-visit interaction as fixed effect, and the study baseline sSE as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p < .0001, Mixed Models Analysis; LSM Difference = 4.361, 95% CI 2-sided [2.220 to 6.501], Standard Error of Mean 1.092
Statistical Analysis 7: Comparison: Placebo vs Lemborexant 5 mg; Month 6 (Statistical analysis 7): Based on MMRM model with factors of age group, region, treatment, visit (Month 6), and treatment-by-visit interaction as fixed effect, and the study baseline sSE as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p = 0.0001, Mixed Models Analysis; LSM Difference = 4.549, 95% CI 2-sided [2.236 to 6.861], Standard Error of Mean 1.179
Statistical Analysis 8: Comparison: Placebo vs Lemborexant 10 mg; Month 6 (Statistical analysis 8): Based on MMRM model with factors of age group, region, treatment, visit (Month 6), and treatment-by-visit interaction as fixed effect, and the study baseline sSE as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p < .0001, Mixed Models Analysis; LSM Difference = 4.667, 95% CI 2-sided [2.373 to 6.960], Standard Error of Mean 1.170

4. Secondary Outcome: Change From Baseline in Subjective Wake After Sleep Onset (sWASO) at the Beginning of Treatment (Mean of the 7 Nights After the First Dose in Placebo-Controlled Period), and at Months 1, 3 and 6
Description: sWASO was defined as sum of estimated minutes of wake during the night after initial sleep onset until the time the participant stopped trying to sleep for the night, operationalized as the time the participant got out of bed for the day.
Time Frame: Baseline, (mean of 7 nights [approximately Week 1]), Months 1, 3 and 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 318 | 316 | 315
minutes
  Baseline: number analyzed (Participants) | 314 | 313 | 311
  Baseline | 132.49 (80.198) | 132.77 (82.518) | 136.83 (87.391)
  Change at first 7 nights: number analyzed (Participants) | 312 | 308 | 309
  Change at first 7 nights | -6.12 (45.893) | -20.21 (46.015) | -23.30 (47.700)
  Change at Month 1: number analyzed (Participants) | 297 | 297 | 293
  Change at Month 1 | -19.01 (50.279) | -23.42 (56.251) | -26.82 (56.989)
  Change at Month 3: number analyzed (Participants) | 278 | 267 | 262
  Change at Month 3 | -27.08 (54.408) | -42.98 (60.064) | -39.42 (62.783)
  Change at Month 6: number analyzed (Participants) | 248 | 244 | 227
  Change at Month 6 | -32.14 (55.279) | -51.45 (67.295) | -48.12 (68.550)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; First 7 nights (Statistical analysis 1): Based on MMRM model with factors of age group, region, treatment, visit (First 7 nights), and treatment-by-visit interaction as fixed effect, and the study baseline sWASO as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p < .0001, Mixed Models Analysis; Least square mean (LSM) Difference = -14.328, 95% CI 2-sided [-21.411 to -7.245], Standard Error of Mean 3.614
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; First 7 nights (Statistical analysis 2): Based on MMRM model with factors of age group, region, treatment, visit (First 7 nights), and treatment-by-visit interaction as fixed effect, and the study baseline sWASO as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p < .0001, Mixed Models Analysis; LSM Difference = -16.720, 95% CI 2-sided [-23.813 to -9.626], Standard Error of Mean 3.619
Statistical Analysis 3: Comparison: Placebo vs Lemborexant 5 mg; Month 1 (Statistical analysis 3): Based on MMRM model with factors of age group, region, treatment, visit (Month 1), and treatment-by-visit interaction as fixed effect, and the study baseline sWASO as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p = 0.1796, Mixed Models Analysis; LSM Difference = -5.514, 95% CI 2-sided [-13.568 to 2.540], Standard Error of Mean 4.109
Statistical Analysis 4: Comparison: Placebo vs Lemborexant 10 mg; Month 1 (Statistical analysis 4): Based on MMRM model with factors of age group, region, treatment, visit (Month 1), and treatment-by-visit interaction as fixed effect, and the study baseline sWASO as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p = 0.0898, Mixed Models Analysis; LSM Difference = -7.005, 95% CI 2-sided [-15.098 to 1.088], Standard Error of Mean 4.129
Statistical Analysis 5: Comparison: Placebo vs Lemborexant 5 mg; Month 3 (Statistical analysis 5): Based on MMRM model with factors of age group, region, treatment, visit (Month 3), and treatment-by-visit interaction as fixed effect, and the study baseline sWASO as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p = 0.0028, Mixed Models Analysis; LSM Difference = -13.424, 95% CI 2-sided [-22.218 to -4.631], Standard Error of Mean 4.486
Statistical Analysis 6: Comparison: Placebo vs Lemborexant 10 mg; Month 3 (Statistical analysis 6): Based on MMRM model with factors of age group, region, treatment, visit (Month 3), and treatment-by-visit interaction as fixed effect, and the study baseline sWASO as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p = 0.0277, Mixed Models Analysis; LSM Difference = -10.079, 95% CI 2-sided [-19.053 to -1.104], Standard Error of Mean 4.578
Statistical Analysis 7: Comparison: Placebo vs Lemborexant 5 mg; Month 6 (Statistical analysis 7): Based on MMRM model with factors of age group, region, treatment, visit (Month 6), and treatment-by-visit interaction as fixed effect, and the study baseline sWASO as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p = 0.0005, Mixed Models Analysis; LSM Difference = -17.474, 95% CI 2-sided [-27.306 to -7.643], Standard Error of Mean 5.014
Statistical Analysis 8: Comparison: Placebo vs Lemborexant 10 mg; Month 6 (Statistical analysis 8): Based on MMRM model with factors of age group, region, treatment, visit (Month 6), and treatment-by-visit interaction as fixed effect, and the study baseline sWASO as a covariate. Missing values are imputed using multiple imputation and assumed to be missing not at random (MNAR/CCMV); Test type: Superiority; p = 0.0105, Mixed Models Analysis; LSM Difference = -12.671, 95% CI 2-sided [-22.378 to -2.964], Standard Error of Mean 4.951

5. Secondary Outcome: Change From Baseline in sTST at the Beginning of Treatment (Mean of the 7 Nights After the First Dose in Placebo-Controlled Period), and at Months 1, 3 and 6
Description: sTST was defined as minutes of sleep from sleep onset to time stopped trying to sleep for the night.
Time Frame: Baseline, (mean of 7 nights [approximately Week 1]), Months 1, 3 and 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 318 | 316 | 315
minutes
  Baseline: number analyzed (Participants) | 307 | 302 | 299
  Baseline | 304.25 (91.459) | 315.52 (93.498) | 306.89 (88.031)
  Change at first 7 nights: number analyzed (Participants) | 303 | 295 | 296
  Change at first 7 nights | 14.78 (54.995) | 34.29 (54.142) | 46.01 (55.110)
  Change at Month 1: number analyzed (Participants) | 291 | 284 | 282
  Change at Month 1 | 30.74 (70.687) | 39.32 (63.548) | 53.22 (67.910)
  Change at Month 3: number analyzed (Participants) | 269 | 256 | 251
  Change at Month 3 | 48.16 (75.859) | 65.82 (71.331) | 70.95 (70.913)
  Change at Month 6: number analyzed (Participants) | 242 | 235 | 220
  Change at Month 6 | 53.53 (74.539) | 76.21 (77.714) | 78.32 (80.741)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; First 7 Nights After the First Dose (Statistical analysis 1): Based on MMRM model with factors of age group, region, treatment, visit (First 7 nights), and treatment-by-visit interaction as fixed effect, and the study baseline sTST as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p < .0001, Mixed Models Analysis; LSM Difference = 22.034, 95% CI 2-sided [13.488 to 30.579], Standard Error of Mean 4.354
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; First 7 nights after the first dose (Statistical analysis 2): Based on MMRM model with factors of age group, region, treatment, visit (First 7 nights), and treatment-by-visit interaction as fixed effect, and the study baseline sTST as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p < .0001, Mixed Models Analysis; LSM Difference = 31.796, 95% CI 2-sided [23.258 to 40.334], Standard Error of Mean 4.350
Statistical Analysis 3: Comparison: Placebo vs Lemborexant 5 mg; Month 1 (Statistical analysis 3): Based on MMRM model with factors of age group, region, treatment, visit (Month 1), and treatment-by-visit interaction as fixed effect, and the study baseline sTST as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.0259, Mixed Models Analysis; LSM Difference = 11.760, 95% CI 2-sided [1.418 to 22.102], Standard Error of Mean 5.269
Statistical Analysis 4: Comparison: Placebo vs Lemborexant 10 mg; Month 1 (Statistical analysis 4): Based on MMRM model with factors of age group, region, treatment, visit (Month 1), and treatment-by-visit interaction as fixed effect, and the study baseline sTST as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p < .0001, Mixed Models Analysis; LSM Difference = 22.131, 95% CI 2-sided [11.757 to 32.505], Standard Error of Mean 5.286
Statistical Analysis 5: Comparison: Placebo vs Lemborexant 5 mg; Month 3 (Statistical analysis 5): Based on MMRM model with factors of age group, region, treatment, visit (Month 3), and treatment-by-visit interaction as fixed effect, and the study baseline sTST as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.0034, Mixed Models Analysis; LSM Difference = 17.374, 95% CI 2-sided [5.781 to 28.968], Standard Error of Mean 5.906
Statistical Analysis 6: Comparison: Placebo vs Lemborexant 10 mg; Month 3 (Statistical analysis 6): Based on MMRM model with factors of age group, region, treatment, visit (Month 3), and treatment-by-visit interaction as fixed effect, and the study baseline sTST as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.0003, Mixed Models Analysis; LSM Difference = 21.686, 95% CI 2-sided [10.014 to 33.359], Standard Error of Mean 5.946
Statistical Analysis 7: Comparison: Placebo vs Lemborexant 5 mg; Month 6 (Statistical analysis 7): Based on MMRM model with factors of age group, region, treatment, visit (Month 6), and treatment-by-visit interaction as fixed effect, and the study baseline sTST as a covariate. Missing values are not imputed and assumed to be missing at random (MAR); Test type: Superiority; p = 0.0034, Mixed Models Analysis; LSM Difference = 18.555, 95% CI 2-sided [6.140 to 30.969], Standard Error of Mean 6.324
Statistical Analysis 8: Comparison: Placebo vs Lemborexant 10 mg; Month 6 (Statistical analysis 8): Based on MMRM model with factors of age group, region, treatment, visit (Month 6), and treatment-by-visit interaction as fixed effect, and the study baseline sTST as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.0004, Mixed Models Analysis; LSM Difference = 22.686, 95% CI 2-sided [10.137 to 35.234], Standard Error of Mean 6.392

6. Secondary Outcome: Percentage of Sleep Onset Responders and Sleep Maintenance Responders at Month 6
Description: Sleep onset responder was defined as follows: sSOL at study Baseline was greater than or equal to (>=) 30 minutes and mean sSOL at 6 months was less than or equal to (<=) 20 minutes. Sleep maintenance responder was defined as follows: sWASO at study Baseline was >=60 minutes and mean sWASO at 6 months was <=60 minutes and showed a reduction of greater than (>)10 minutes compared to Study Baseline.
Time Frame: Month 6
Population: The FAS was the group of randomized participants who received at least one dose of randomized study drug and had at least one postdose primary efficacy measurement. Number analyzed refers to number of participants evaluable for specified category.
Measure: Number; unit: percentage of responders
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 318 | 316 | 315
percentage of responders
  Sleep Onset Responders: number analyzed (Participants) | 254 | 250 | 249
  Sleep Onset Responders | 17.7 | 31.2 | 30.1
  Sleep Maintenance Responders: number analyzed (Participants) | 250 | 263 | 257
  Sleep Maintenance Responders | 20.4 | 35.0 | 30.0
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; Sleep onset responders: Statistical analysis 1; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel; Difference of percentage = 13.67, 95% CI 2-sided [6.24 to 21.10]
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; Sleep Onset Responders: Statistical analysis 2; Test type: Superiority; p = 0.0009, Cochran-Mantel-Haenszel; Difference of percentage = 12.53, 95% CI 2-sided [5.20 to 19.86]
Statistical Analysis 3: Comparison: Placebo vs Lemborexant 5 mg; Sleep Maintenance Responders: Statistical analysis 3; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Difference of percentage = 14.65, 95% CI 2-sided [6.97 to 22.33]
Statistical Analysis 4: Comparison: Placebo vs Lemborexant 10 mg; Sleep Maintenance Responders: Statistical analysis 4; Test type: Superiority; p = 0.0110, Cochran-Mantel-Haenszel; Difference of percentage = 9.82, 95% CI 2-sided [2.29 to 17.35]

7. Secondary Outcome: Percentage of Sleep Onset Responders and Sleep Maintenance Responders at Month 12
Description: Sleep onset responder was defined as follows: sSOL at study Baseline was >=30 minutes and mean sSOL at 6 months was <=20 minutes. Sleep maintenance responder was defined as follows: sWASO at study Baseline was >=60 minutes and mean sWASO at 6 months was <=60 minutes and showed a reduction of > 10 minutes compared to study Baseline.
Time Frame: Month 12
Population: Overall participants analyzed based on number in "On-Treatment FAS (Participants who received at least 1 dose of lemborexant and had at least 1 postdose primary efficacy measurement)". Hence, these numbers include lemborexant data from participants re-randomized from placebo in Period 1. Number analyzed=participants analyzed at specified timepoint.
Measure: Number; unit: percentage of participants
Groups:
- Lemborexant 5 mg: Participants received lemborexant 5 mg/placebo, tablets, orally, once daily through Month 1-6 (in Period 1) and lemborexant 5 mg, tablets, orally, once daily through Month 7-12 (in Period 2).
- Lemborexant 10 mg: Participants received lemborexant 10 mg/placebo, tablets, orally, once daily through Month 1-6 (in Period 1) and lemborexant 10 mg, tablets, orally, once daily through Month 7-12 (in Period 2).
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 444 | 437
percentage of participants
  Sleep Onset Responders: number analyzed (Participants) | 310 | 285
  Sleep Onset Responders | 34.2 | 37.2
  Sleep Maintainance Responders: number analyzed (Participants) | 317 | 280
  Sleep Maintainance Responders | 35.0 | 39.6

8. Secondary Outcome: Change From Baseline in Insomnia Severity Index (ISI) Daytime Functioning Score at Months 1, 3, and 6
Description: The ISI is a 4-7 item, self-report questionnaire assessing the nature, severity, and impact of insomnia. The dimensions evaluated were: 1. severity of sleep onset; 2. sleep maintenance; 3. early morning awakening problems; 4. sleep dissatisfaction; 5. interference of sleep difficulties with daytime functioning; 6. noticeability of the sleep problems by others; and 7. distress caused by the sleep difficulties. A 5-point Likert scale was used to rate each item (from 0=no problem to 4=very severe problem). Daytime functioning score (sum of items 4 to 7) were analyzed. Higher score indicated severe insomnia problem. The total score range for sum of items is 0-16.
Time Frame: Baseline, Months 1, 3, and 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Participants received lemborexant-matched placebo, tablet, orally, once daily for up to Month 6 in the placebo-controlled treatment period. Then they were re-randomized to Lemborexant 5 mg or Lemborexant 10 mg.
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 318 | 316 | 315
score on a scale
  Baseline | 11.0 (2.10) | 11.4 (2.02) | 11.0 (2.15)
  Change at Month 1: number analyzed (Participants) | 296 | 300 | 286
  Change at Month 1 | -3.1 (3.41) | -4.1 (3.66) | -4.2 (4.01)
  Change at Month 3: number analyzed (Participants) | 283 | 274 | 259
  Change at Month 3 | -3.7 (3.55) | -5.2 (3.88) | -5.2 (4.05)
  Change at Month 6: number analyzed (Participants) | 257 | 258 | 234
  Change at Month 6 | -4.3 (3.66) | -6.0 (3.76) | -5.7 (4.00)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; Month 1 (Statistical analysis 1): Based on MMRM model with factors for age group, region, treatment, visit (Month 1), and treatment-by-visit interaction as fixed effects, and study baseline ISI score as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.0137, Mixed Models Analysis; LSM Difference = -0.71, 95% CI 2-sided [-1.27 to -0.15], Standard Error of Mean 0.287
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; Month 1 (Statistical analysis 2): Based on MMRM model with factors for age group, region, treatment, visit (Month 1), and treatment-by-visit interaction as fixed effects, and study baseline ISI score as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.0011, Mixed Models Analysis; LSM Difference = -0.94, 95% CI 2-sided [-1.51 to -0.38], Standard Error of Mean 0.289
Statistical Analysis 3: Comparison: Placebo vs Lemborexant 5 mg; Month 3 (Statistical analysis 3): Based on MMRM model with factors for age group, region, treatment, visit (Month 3), and treatment-by-visit interaction as fixed effects, and study baseline ISI score as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.0001, Mixed Models Analysis; LSM Difference = -1.16, 95% CI 2-sided [-1.75 to -0.57], Standard Error of Mean 0.302
Statistical Analysis 4: Comparison: Placebo vs Lemborexant 10 mg; Month 3 (Statistical analysis 4): Based on MMRM model with factors for age group, region, treatment, visit (Month 3), and treatment-by-visit interaction as fixed effects, and study baseline ISI score as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p < .0001, Mixed Models Analysis; LSM Difference = -1.36, 95% CI 2-sided [-1.96 to -0.76], Standard Error of Mean 0.305
Statistical Analysis 5: Comparison: Placebo vs Lemborexant 5 mg; Month 6 (Statistical analysis 5): Based on MMRM model with factors for age group, region, treatment, visit (Month 6), and treatment-by-visit interaction as fixed effects, and study baseline ISI score as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p < .0001, Mixed Models Analysis; LSM Difference = -1.30, 95% CI 2-sided [-1.90 to -0.71], Standard Error of Mean 0.302
Statistical Analysis 6: Comparison: Placebo vs Lemborexant 10 mg; Month 6 (Statistical analysis 6): Based on MMRM model with factors for age group, region, treatment, visit (Month 6), and treatment-by-visit interaction as fixed effects, and study baseline ISI score as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p < .0001, Mixed Models Analysis; LSM Difference = -1.32, 95% CI 2-sided [-1.92 to -0.71], Standard Error of Mean 0.307

9. Secondary Outcome: Change From Baseline in Fatigue Severity Scale (FSS) Total Score at Months 1, 3 and 6
Description: The FSS is a self-reported scale on which participants were instructed to choose a number from 1 to 7 that indicated their degree of agreement with 9 statements about their fatigue where "1" indicates strongly disagree and "7", strongly agree. The FSS total score was the sum of all responses to the 9 questions. Higher total scores and average item scores indicated greater fatigue. Total score range is 9 to 63.
Time Frame: Baseline, Months 1, 3 and 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 318 | 316 | 315
score on a scale
  Baseline | 35.2 (13.55) | 37.4 (12.74) | 36.0 (13.01)
  Change at Month 1: number analyzed (Participants) | 296 | 300 | 286
  Change at Month 1 | -3.9 (11.62) | -6.6 (11.83) | -6.4 (13.68)
  Change at Month 3: number analyzed (Participants) | 283 | 274 | 259
  Change at Month 3 | -4.3 (11.37) | -7.7 (12.97) | -7.9 (13.56)
  Change at Month 6: number analyzed (Participants) | 257 | 258 | 234
  Change at Month 6 | -6.3 (12.07) | -10.1 (13.56) | -8.9 (14.91)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; Month 1 (Statistical analysis 1): Based on MMRM model with factors for age group, region, treatment, visit (Month 1), and treatment-by-visit interaction as fixed effects, and study baseline FSS score as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.0670, Mixed Models Analysis; LSM Difference = -1.66, 95% CI 2-sided [-3.44 to 0.12], Standard Error of Mean 0.905
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; Month 1 (Statistical analysis 2): Based on MMRM model with factors for age group, region, treatment, visit (Month 1), and treatment-by-visit interaction as fixed effects, and study baseline FSS score as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.0257, Mixed Models Analysis; LSM Difference = -2.04, 95% CI 2-sided [-3.83 to -0.25], Standard Error of Mean 0.913
Statistical Analysis 3: Comparison: Placebo vs Lemborexant 5 mg; Month 3 (Statistical analysis 3): Based on MMRM model with factors for age group, region, treatment, visit (Month 3), and treatment-by-visit interaction as fixed effects, and study baseline FSS score as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.0206, Mixed Models Analysis; LSM Difference = -2.18, 95% CI 2-sided [-4.02 to -0.34], Standard Error of Mean 0.939
Statistical Analysis 4: Comparison: Placebo vs Lemborexant 10 mg; Month 3 (Statistical analysis 4): Based on MMRM model with factors for age group, region, treatment, visit (Month 3), and treatment-by-visit interaction as fixed effects, and study baseline FSS score as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.0014, Mixed Models Analysis; LSM Difference = -3.04, 95% CI 2-sided [-4.91 to -1.18], Standard Error of Mean 0.950
Statistical Analysis 5: Comparison: Placebo vs Lemborexant 5 mg; Month 6 (Statistical analysis 5): Based on MMRM model with factors for age group, region, treatment, visit (Month 6), and treatment-by-visit interaction as fixed effects, and study baseline FSS score as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.0134, Mixed Models Analysis; LSM Difference = -2.50, 95% CI 2-sided [-4.48 to -0.52], Standard Error of Mean 0.112
Statistical Analysis 6: Comparison: Placebo vs Lemborexant 10 mg; Month 6 (Statistical analysis 6): Based on MMRM model with factors for age group, region, treatment, visit (Month 6), and treatment-by-visit interaction as fixed effects, and study baseline FSS score as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.0128, Mixed Models Analysis; LSM Difference = -2.56, 95% CI 2-sided [-4.57 to -0.54], Standard Error of Mean 1.026

10. Secondary Outcome: Change From Baseline in Mean Rating on the Morning Sleepiness Item of the Sleep Diary at the Beginning of Treatment (Mean of the 7 Nights After the First Dose in Placebo-Controlled Period), and at Months 1, 3 and 6
Description: The Sleep Diary was used to assess subjective ratings of morning sleepiness with the following question:
  "How sleepy/alert do you feel this morning?" Participants rated their sleepiness/alertness level on a scale from 1 to 9, with 1 being extremely poor (sleepy) and 9 being extremely good (alert). Higher score indicated better outcome.
Time Frame: Baseline, (mean of 7 nights [approximately Week 1]) in placebo-controlled period, Month 1, 3, 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 318 | 316 | 315
score on a scale
  Baseline: number analyzed (Participants) | 316 | 314 | 312
  Baseline | 3.94 (1.558) | 3.93 (1.349) | 3.93 (1.324)
  Change at First 7 nights: number analyzed (Participants) | 314 | 310 | 310
  Change at First 7 nights | 0.15 (0.991) | 0.36 (0.964) | 0.33 (1.018)
  Change at Month 1: number analyzed (Participants) | 300 | 298 | 297
  Change at Month 1 | 0.44 (1.233) | 0.53 (1.172) | 0.55 (1.298)
  Change at Month 3: number analyzed (Participants) | 280 | 268 | 264
  Change at Month 3 | 0.62 (1.366) | 0.74 (1.325) | 0.90 (1.452)
  Change at Month 6: number analyzed (Participants) | 249 | 245 | 229
  Change at Month 6 | 0.79 (1.392) | 0.98 (1.463) | 1.05 (1.524)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; First 7 nights (Statistical analysis): Based on MMRM model with factors of age group, region, treatment, visit (First 7 nights), and treatment-by-visit interaction as fixed effect, and the study baseline Mean Rating on Morning Sleepiness as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.0067, Mixed Models Analysis; LSM Difference = 0.205, 95% CI 2-sided [0.057 to 0.353], Standard Error of Mean 0.076
Statistical Analysis 2: Comparison: Placebo vs Lemborexant 10 mg; First 7 nights (Statistical analysis 2): Based on MMRM model with factors of age group, region, treatment, visit (First 7 nights), and treatment-by-visit interaction as fixed effect, and the study baseline Mean Rating on Morning Sleepiness as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.0237, Mixed Models Analysis; LSM Difference = 0.171, 95% CI 2-sided [0.023 to 0.320], Standard Error of Mean 0.076
Statistical Analysis 3: Comparison: Placebo vs Lemborexant 5 mg; Month 1 (Statistical analysis 3): Based on MMRM model with factors of age group, region, treatment, visit (Month 1), and treatment-by-visit interaction as fixed effect, and the study baseline Mean Rating on Morning Sleepiness as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.4120, Mixed Models Analysis; LSM Difference = 0.077, 95% CI 2-sided [-0.107 to 0.261], Standard Error of Mean 0.094
Statistical Analysis 4: Comparison: Placebo vs Lemborexant 10 mg; Month 1 (Statistical analysis 4): Based on MMRM model with factors of age group, region, treatment, visit (Month 1), and treatment-by-visit interaction as fixed effect, and the study baseline Mean Rating on Morning Sleepiness as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.4347, Mixed Models Analysis; LSM Difference = 0.073, 95% CI 2-sided [-0.111 to 0.258], Standard Error of Mean 0.094
Statistical Analysis 5: Comparison: Placebo vs Lemborexant 5 mg; Month 3 (Statistical analysis 5): Based on MMRM model with factors of age group, region, treatment, visit (Month 3), and treatment-by-visit interaction as fixed effect, and the study baseline Mean Rating on Morning Sleepiness as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.4992, Mixed Models Analysis; LSM Difference = 0.074, 95% CI 2-sided [-0.141 to 0.289], Standard Error of Mean 0.109
Statistical Analysis 6: Comparison: Placebo vs Lemborexant 10 mg; Month 3 (Statistical analysis 6): Based on MMRM model with factors of age group, region, treatment, visit (Month 3), and treatment-by-visit interaction as fixed effect, and the study baseline Mean Rating on Morning Sleepiness as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.0208, Mixed Models Analysis; LSM Difference = 0.255, 95% CI 2-sided [0.039 to 0.471], Standard Error of Mean 0.110
Statistical Analysis 7: Comparison: Placebo vs Lemborexant 5 mg; Month 6 (Statistical analysis 7): Based on MMRM model with factors of age group, region, treatment, visit (Month 6), and treatment-by-visit interaction as fixed effect, and the study baseline Mean Rating on Morning Sleepiness as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.2248, Mixed Models Analysis; LSM Difference = 0.144, 95% CI 2-sided [-0.089 to 0.378], Standard Error of Mean 0.119
Statistical Analysis 8: Comparison: Placebo vs Lemborexant 10 mg; Month 6 (Statistical analysis 8): Based on MMRM model with factors of age group, region, treatment, visit (Month 6), and treatment-by-visit interaction as fixed effect, and the study baseline Mean Rating on Morning Sleepiness as a covariate. Missing values are not imputed and assumed to be MAR; Test type: Superiority; p = 0.0298, Mixed Models Analysis; LSM Difference = 0.261, 95% CI 2-sided [0.026 to 0.497], Standard Error of Mean 0.120

11. Secondary Outcome: Change From Baseline in Mean Rating on the Morning Sleepiness Item of the Sleep Diary at the Beginning of Treatment (Mean of the 7 Nights After the First Dose in Active Treatment Period)
Time Frame: Baseline, First 7 nights (approximately Week 1) in active treatment period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 444 | 437
score on a scale
  Baseline: number analyzed (Participants) | 442 | 434
  Baseline | 4.15 (1.516) | 4.16 (1.428)
  Change at First 7 nights: number analyzed (Participants) | 310 | 310
  Change at First 7 nights | 0.36 (0.964) | 0.33 (1.018)

12. Secondary Outcome: Change From Screening in Mean Rating on the Morning Sleepiness Item of the Sleep Diary at the First and Second 7 Mornings of the Follow-up Period
Description: as for outcome 10
Time Frame: Screening, First and second 7 mornings in follow-up period (Week 52 to 54)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 444 | 437
score on a scale
  Screening: number analyzed (Participants) | 440 | 436
  Screening | 3.63 (1.393) | 3.54 (1.197)
  Change at First 7 mornings: number analyzed (Participants) | 335 | 328
  Change at First 7 mornings | 1.03 (1.615) | 1.32 (1.611)
  Change at Second 7 mornings: number analyzed (Participants) | 327 | 313
  Change at Second 7 mornings | 0.98 (1.699) | 1.22 (1.635)

13. Secondary Outcome: Change From Baseline in Mean Rating on the Morning Sleepiness Item of the Sleep Diary at Months 1, 3, 6, 9 and 12
Description: as for outcome 10
Time Frame: Baseline, Months 1, 3, 6, 9 and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 444 | 437
score on a scale
  Baseline: number analyzed (Participants) | 442 | 434
  Baseline | 4.15 (1.516) | 4.16 (1.428)
  Change at Month 1 of exposure: number analyzed (Participants) | 415 | 412
  Change at Month 1 of exposure | 0.46 (1.082) | 0.42 (1.223)
  Change at Month 3 of exposure: number analyzed (Participants) | 386 | 375
  Change at Month 3 of exposure | 0.60 (1.264) | 0.70 (1.356)
  Change at Month 6 of exposure: number analyzed (Participants) | 352 | 331
  Change at Month 6 of exposure | 0.78 (1.424) | 0.86 (1.461)
  Change at Month 9 of exposure: number analyzed (Participants) | 233 | 213
  Change at Month 9 of exposure | 1.00 (1.512) | 1.08 (1.489)
  Change at Month 12 of exposure: number analyzed (Participants) | 216 | 204
  Change at Month 12 of exposure | 1.11 (1.499) | 1.31 (1.604)

14. Secondary Outcome: Rebound Insomnia: Mean sSOL on Each of the First 3 Nights, First 7 Nights, and Last 7 Nights of the Follow-up Period
Description: Rebound Insomnia: Rebound insomnia was defined as insomnia that occurred following discontinuation of a sedative substance taken to relieve primary insomnia. sSOL was defined as estimated minutes from the time that the participant attempted to sleep until sleep onset.
Time Frame: First 3 nights, first and Last 7 nights of the follow up period (Week 52 to 54)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 444 | 437
minutes
  Mean of first 3 nights: number analyzed (Participants) | 287 | 284
  Mean of first 3 nights | 40.35 (48.661) | 41.73 (55.694)
  Mean sSOL of the first 7 nights: number analyzed (Participants) | 337 | 328
  Mean sSOL of the first 7 nights | 41.35 (38.967) | 41.90 (47.826)
  Mean sSOL of the second 7 nights: number analyzed (Participants) | 329 | 312
  Mean sSOL of the second 7 nights | 44.10 (38.030) | 41.30 (47.471)

15. Secondary Outcome: Rebound Insomnia: Mean sWASO on Each of the First 3 Nights, First 7 Nights, and Last 7 Nights of the Follow-up Period
Description: Rebound Insomnia: Rebound insomnia was defined as insomnia that occurred following discontinuation of a sedative substance taken to relieve primary insomnia. sWASO was defined as sum of estimated minutes of wake during the night after initial sleep onset until the time the participant stopped trying to sleep for the night, operationalized as the time the participant got out of bed for the day.
Time Frame: First 3 nights, first and last 7 nights of the follow up period (Week 52 to 54)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 444 | 437
minutes
  Mean of first 3 nights: number analyzed (Participants) | 282 | 282
  Mean of first 3 nights | 86.66 (80.038) | 97.88 (83.302)
  Mean of the first 7 nights: number analyzed (Participants) | 337 | 326
  Mean of the first 7 nights | 91.56 (81.738) | 95.79 (79.784)
  Mean of the Last 7 nights: number analyzed (Participants) | 329 | 312
  Mean of the Last 7 nights | 92.62 (82.672) | 98.19 (80.668)

16. Secondary Outcome: Rebound Insomnia: Percentage of Participants Whose sSOL Was Longer Than at Screening for First 3 Nights of the Follow-up Period, or Whom Mean sSOL Was Longer Than at Screening for First 7 Nights or Last 7 Nights of the Follow-up Period
Description: as for outcome 14
Time Frame: First 3 nights, first and last 7 nights of the follow up period (Week 52 to 54)
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 444 | 437
percentage of participants
  Average of first 3 nights: number analyzed (Participants) | 285 | 284
  Average of first 3 nights | 9.46 | 9.38
  Average of first 7 nights: number analyzed (Participants) | 335 | 328
  Average of first 7 nights | 11.94 | 10.53
  Average of second 7 nights: number analyzed (Participants) | 327 | 312
  Average of second 7 nights | 11.71 | 9.38

17. Secondary Outcome: Rebound Insomnia: Percentage of Participants Whose sWASO is Higher Than at Screening for First 3 Nights of the Follow-up Period, or Whose Mean sWASO is Higher Than at Screening for the First 7 Nights or Last 7 Nights of the Follow-up Period
Description: as for outcome 15
Time Frame: First 3 nights, First and Last 7 nights of the follow up period (Week 52 to 54)
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 444 | 437
percentage of participants
  Average of first 3 nights: number analyzed (Participants) | 280 | 282
  Average of first 3 nights | 11.26 | 12.59
  Average of first 7 nights: number analyzed (Participants) | 335 | 325
  Average of first 7 nights | 12.39 | 14.19
  Average of second 7 nights: number analyzed (Participants) | 327 | 311
  Average of second 7 nights | 13.51 | 11.90

18. Secondary Outcome: Persistence of Effect: Mean Change From Baseline in sSOL, sWASO, and sTST at Months 3, 6, 9, and 12 Compared to Month 1
Description: sSOL was defined as estimated minutes from the time that the participant attempted to sleep until sleep onset. sWASO was defined as sum of estimated minutes of wake during the night after initial sleep onset until the time the participant stopped trying to sleep for the night, operationalized as the time the participant got out of bed for the day. sTST: minutes of sleep from sleep onset to time stopped trying to sleep for the night. At each month beyond Month 1, the change from Baseline was compared to either the lower bound of the 95% CI (for sTST) or the upper bound of the 95% CI (for sSOL and sWASO) at Month 1. Persistence of efficacy was defined as present if the mean change from Baseline at Month 6 was above the lower bound of the 95% CI at Month 1 for sTST and below the upper bound of the 95% CI at Month 1 for sSOL and sWASO.
Time Frame: Baseline, Month 1, 3, 6, 9, 12
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 444 | 437
minutes
  sSOL: Change at Month 1 of exposure: number analyzed (Participants) | 415 | 412
  sSOL: Change at Month 1 of exposure | -17.17 [-19.76 to -14.58] | -18.64 [-21.26 to -16.02]
  sSOL: Change at Month 3 of exposure: number analyzed (Participants) | 386 | 375
  sSOL: Change at Month 3 of exposure | -21.47 [-24.46 to -18.48] | -21.58 [-24.61 to -18.54]
  sSOL: Change at Month 6 of exposure: number analyzed (Participants) | 352 | 331
  sSOL: Change at Month 6 of exposure | -24.13 [-27.22 to -21.04] | -22.99 [-26.14 to -19.83]
  sSOL: Change at Month 9 of exposure: number analyzed (Participants) | 233 | 213
  sSOL: Change at Month 9 of exposure | -26.00 [-29.25 to -22.75] | -27.36 [-30.70 to -24.01]
  sSOL: Change at Month 12 of exposure: number analyzed (Participants) | 216 | 214
  sSOL: Change at Month 12 of exposure | -25.83 [-29.44 to -22.22] | -26.32 [-30.03 to -22.61]
  sWASO: Change at Month 1 of exposure: number analyzed (Participants) | 414 | 408
  sWASO: Change at Month 1 of exposure | -17.26 [-22.54 to -11.97] | -18.69 [-24.05 to -13.33]
  sWASO: Change at Month 3 of exposure: number analyzed (Participants) | 385 | 373
  sWASO: Change at Month 3 of exposure | -31.34 [-37.12 to -25.57] | -28.97 [-34.86 to -23.09]
  sWASO: Change at Month 6 of exposure: number analyzed (Participants) | 351 | 329
  sWASO: Change at Month 6 of exposure | -36.10 [-42.57 to -29.63] | -31.54 [-38.16 to -24.91]
  sWASO: Change at Month 9 of exposure: number analyzed (Participants) | 232 | 212
  sWASO: Change at Month 9 of exposure | -39.28 [-46.74 to -31.83] | -40.39 [-48.08 to -32.71]
  sWASO: Change at Month 12 of exposure: number analyzed (Participants) | 215 | 203
  sWASO: Change at Month 12 of exposure | -42.87 [-50.13 to -35.61] | -43.76 [-51.21 to -36.31]
  sTST: Change at Month 1 of exposure: number analyzed (Participants) | 400 | 396
  sTST: Change at Month 1 of exposure | 31.98 [25.54 to 38.42] | 38.04 [31.51 to 44.57]
  sTST: Change at Month 3 of exposure: number analyzed (Participants) | 373 | 361
  sTST: Change at Month 3 of exposure | 49.27 [42.33 to 56.22] | 53.51 [46.42 to 60.61]
  sTST: Change at Month 6 of exposure: number analyzed (Participants) | 342 | 321
  sTST: Change at Month 6 of exposure | 54.99 [47.18 to 62.80] | 56.36 [48.35 to 64.36]
  sTST: Change at Month 9 of exposure: number analyzed (Participants) | 222 | 205
  sTST: Change at Month 9 of exposure | 55.41 [46.49 to 64.33] | 61.13 [51.93 to 70.32]
  sTST: Change at Month 12 of exposure: number analyzed (Participants) | 207 | 196
  sTST: Change at Month 12 of exposure | 58.15 [49.29 to 67.01] | 66.50 [57.41 to 75.60]

19. Secondary Outcome: Persistence of Effect: Mean Change From Baseline in sSE at Months 3, 6, 9, and 12 Compared to Month 1
Description: sSE was defined as percentage of sTST per subjective time spent in bed, calculated as the interval from the time the participant reports attempting to sleep until the time the participant stopped trying to sleep for the night (operationalized as the time the participant got out of bed for the day), and time spent asleep derived from subjective time spent in bed minus sWASO. At each month beyond Month 1, the change from Baseline was compared to the lower bound of the 95% CI at Month 1. Persistence of efficacy was defined as present if the mean change from Baseline at Month 6 was above the lower bound of the 95% CI at Month 1 for sSE.
Time Frame: Baseline, Months 1, 3, 6, 9, and 12
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of sTST
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 444 | 437
percentage of sTST
  Change at Month 1 of exposure: number analyzed (Participants) | 400 | 396
  Change at Month 1 of exposure | 6.35 [5.13 to 7.57] | 7.32 [6.09 to 8.56]
  Change at Month 3 of exposure: number analyzed (Participants) | 373 | 361
  Change at Month 3 of exposure | 10.01 [8.69 to 11.34] | 10.25 [8.90 to 11.60]
  Change at Month 6 of exposure: number analyzed (Participants) | 342 | 321
  Change at Month 6 of exposure | 11.10 [9.61 to 12.58] | 11.08 [9.56 to 12.60]
  Change at Month 9 of exposure: number analyzed (Participants) | 222 | 205
  Change at Month 9 of exposure | 11.85 [10.13 to 13.56] | 12.84 [11.08 to 14.61]
  Change at Month 12 of exposure: number analyzed (Participants) | 207 | 196
  Change at Month 12 of exposure | 12.61 [10.92 to 14.31] | 13.66 [11.92 to 15.40]

20. Secondary Outcome: Persistence of Effect: Mean Change From Period 2 Baseline (Month 6) in sSOL, sWASO, and sTST at Months 9 and 12 Compared to Month 7
Description: sSOL is defined as estimated minutes from the time that the participant attempted to sleep until sleep onset. sWASO: sum of estimated minutes of wake during the night after initial sleep onset until the time the participant stopped trying to sleep for the night, operationalized as the time the participant got out of bed for the day. sTST: minutes of sleep from sleep onset to time stopped trying to sleep for the night. At each month beyond Month 7, the change from Baseline was compared to either the lower bound of the 95% CI for sTST or the upper bound of the 95% CI (for sSOL and sWASO) at Month 7. Persistence of effect was defined as present if the mean change from Baseline at Month 12 was above the lower bound of the 95% CI at Month 7 for sTST and below the upper bound of the 95% CI at Month 7 for sSOL and sWASO.
Time Frame: Baseline, Month 7, 9, 12
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 444 | 437
minutes
  sSOL: Change at Month 7 of exposure: number analyzed (Participants) | 355 | 334
  sSOL: Change at Month 7 of exposure | -28.55 [-32.39 to -24.70] | -29.46 [-33.42 to -25.50]
  sSOL: Change at Month 9 of exposure: number analyzed (Participants) | 349 | 324
  sSOL: Change at Month 9 of exposure | -32.10 [-35.39 to -28.80] | -30.91 [-34.31 to -27.52]
  sSOL: Change at Month 12 of exposure: number analyzed (Participants) | 323 | 306
  sSOL: Change at Month 12 of exposure | -31.40 [-34.85 to -27.96] | -31.33 [-34.88 to -27.78]
  sWASO: Change at Month 7 of exposure: number analyzed (Participants) | 355 | 334
  sWASO: Change at Month 7 of exposure | -45.62 [-52.53 to -38.70] | -43.09 [-50.20 to -35.99]
  sWASO: Change at Month 9 of exposure: number analyzed (Participants) | 349 | 324
  sWASO: Change at Month 9 of exposure | -47.70 [-54.54 to -40.86] | -48.87 [-55.92 to -41.82]
  sWASO: Change at Month 12 of exposure: number analyzed (Participants) | 323 | 306
  sWASO: Change at Month 12 of exposure | -48.46 [-55.35 to -41.57] | -49.28 [-56.36 to -42.19]
  sTST: Change at Month 7 of exposure: number analyzed (Participants) | 355 | 334
  sTST: Change at Month 7 of exposure | 75.00 [65.30 to 84.71] | 76.95 [66.97 to 86.92]
  sTST: Change at Month 9 of exposure: number analyzed (Participants) | 349 | 324
  sTST: Change at Month 9 of exposure | 78.69 [68.99 to 88.39] | 81.24 [71.26 to 91.23]
  sTST: Change at Month 12 of exposure: number analyzed (Participants) | 323 | 306
  sTST: Change at Month 12 of exposure | 78.61 [68.61 to 88.61] | 83.61 [73.33 to 93.90]

21. Secondary Outcome: Persistence of Effect: Mean Change From Period 2 Baseline (Month 6) in sSE at Months 9 and 12 Compared to Month 7
Description: sSE: percentage of sTST per subjective time spent in bed, calculated as the interval from the time the participant reports attempting to sleep until the time the participant stopped trying to sleep for the night (operationalized as the time the subject got out of bed for the day), and time spent asleep derived from subjective time spent in bed minus sWASO. At each month beyond Month 7, the change from Baseline was compared to the lower bound of the 95% CI for sSE at Month 7. Persistence of effect was defined as present if the mean change from Baseline at Month 12 was above the lower bound of the 95% CI at Month 7 for sSE.
Time Frame: Baseline, Month 7, 9, 12
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of sTST
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 444 | 437
percentage of sTST
  Change at Month 7 of exposure: number analyzed (Participants) | 354 | 334
  Change at Month 7 of exposure | 12.88 [9.01 to 16.75] | 15.12 [11.13 to 19.10]
  Change at Month 9 of exposure: number analyzed (Participants) | 349 | 324
  Change at Month 9 of exposure | 16.54 [14.88 to 18.20] | 16.49 [14.78 to 18.20]
  Change at Month 12 of exposure: number analyzed (Participants) | 323 | 306
  Change at Month 12 of exposure | 16.34 [14.70 to 17.98] | 16.82 [15.13 to 18.50]

22. Secondary Outcome: Persistence of Effect: Mean Change From Study Baseline and Period 2 Baseline (Month 6) in sSOL, sWASO, and sTST at Months 3 and 6 Exposure Compared to Month 1
Description: sSOL was defined as estimated minutes from the time that the participant attempted to sleep until sleep onset. sWASO: sum of estimated minutes of wake during the night after initial sleep onset until the time the participant stopped trying to sleep for the night, operationalized as the time the participant got out of bed for the day. sTST: minutes of sleep from sleep onset to time stopped trying to sleep for the night. At 3 and 6 months of exposure, the change from Baseline was compared to either the lower bound of the 95% CI for sTST or the upper bound of the 95% CI (for sSOL and sWASO) at 1 month of exposure. Persistence of effect was defined as present if the mean change from Baseline at 6 months of exposure was above the lower bound of the 95% CI at 1 month of exposure for sTST and below the upper bound of the 95% CI at 1 month of exposure for sSOL and sWASO.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 444 | 437
minutes
  sSOL: Change at Month 1 of exposure: number analyzed (Participants) | 415 | 412
  sSOL: Change at Month 1 of exposure | -17.17 [-19.76 to -14.58] | -18.64 [-21.26 to -16.02]
  sSOL: Change at Month 3 of exposure: number analyzed (Participants) | 386 | 375
  sSOL: Change at Month 3 of exposure | -21.47 [-24.46 to -18.48] | -21.58 [-24.61 to -18.54]
  sSOL: Change at Month 6 of exposure: number analyzed (Participants) | 352 | 331
  sSOL: Change at Month 6 of exposure | -24.13 [-27.22 to -21.04] | -22.99 [-26.14 to -19.83]
  sWASO: Change at Month 1 of exposure: number analyzed (Participants) | 414 | 408
  sWASO: Change at Month 1 of exposure | -17.26 [-22.54 to -11.97] | -18.69 [-24.05 to -13.33]
  sWASO: Change at Month 3 of exposure: number analyzed (Participants) | 385 | 373
  sWASO: Change at Month 3 of exposure | -31.34 [-37.12 to -25.57] | -28.97 [-34.86 to -23.09]
  sWASO: Change at Month 6 of exposure: number analyzed (Participants) | 351 | 329
  sWASO: Change at Month 6 of exposure | -36.10 [-42.57 to -29.63] | -31.54 [-38.16 to -24.91]
  sTST: Change at Month 1 of exposure: number analyzed (Participants) | 400 | 396
  sTST: Change at Month 1 of exposure | 31.98 [25.54 to 38.42] | 38.04 [31.51 to 44.57]
  sTST: Change at Month 3 of exposure: number analyzed (Participants) | 373 | 361
  sTST: Change at Month 3 of exposure | 49.27 [42.33 to 56.22] | 53.51 [46.42 to 60.61]
  sTST: Change at Month 6 of exposure: number analyzed (Participants) | 342 | 321
  sTST: Change at Month 6 of exposure | 54.99 [47.18 to 62.80] | 56.36 [48.35 to 64.36]

23. Secondary Outcome: Persistence of Effect: Mean Change From Study Baseline and Period 2 Baseline (Month 6) in sSE at Months 3 and 6 Exposure Compared to Month 1
Description: sSE was defined as percentage of sTST per subjective time spent in bed, calculated as the interval from the time the participant reports attempting to sleep until the time the participant stopped trying to sleep for the night (operationalized as the time the participant got out of bed for the day), and time spent asleep derived from subjective time spent in bed minus sWASO. At 3 and 6 months of exposure, the change from Baseline was compared to the lower bound of the 95% CI for sSE at 1 month of exposure. Persistence of effect was defined as present if the mean change from Baseline at 6 months of exposure was above the lower bound of the 95% CI at 1 month of exposure for sSE.
Time Frame: Baseline, Month 1, 3, 6
Population: On-treatment FAS was the group of participants who received at least 1 dose of lemborexant and had at least 1 post dose primary efficacy measurement. Overall Participants Analyzed here is based on the number in the "On-Treatment FAS". Hence these numbers include the lemborexant data from the participants re-randomized from placebo in Period 1.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of sTST
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 444 | 437
percentage of sTST
  Change at Month 1 of exposure: number analyzed (Participants) | 400 | 396
  Change at Month 1 of exposure | 6.35 [5.13 to 7.57] | 7.32 [6.09 to 8.56]
  Change at Month 3 of exposure: number analyzed (Participants) | 373 | 361
  Change at Month 3 of exposure | 10.01 [8.69 to 11.34] | 10.25 [8.90 to 11.60]
  Change at Month 6 of exposure: number analyzed (Participants) | 342 | 321
  Change at Month 6 of exposure | 11.10 [9.61 to 12.58] | 11.08 [9.56 to 12.60]

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Week 54
Description: Placebo arm included AE data for participants who received placebo in Period 1. Lemborexant 5 mg and 10 mg arms included AE data of participants who received either lemborexant 5 mg or 10 mg throughout the study (Period 1 and 2 both) and participants re-randomized from placebo (in Period 1) to either lemborexant 5 mg or lemborexant 10 mg in Period 2.
Groups:
- Placebo: Participants received placebo matched to lemborexant tablet, orally, once daily for up to 6 months. Then they were re-randomized to Lemborexant 5 mg or Lemborexant 10 mg.
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
All-Cause Mortality (participants affected / at risk) | 0/319 | 0/447 | 0/437
Serious Adverse Events (participants affected / at risk) | 5/319 | 18/447 | 16/437
Other Adverse Events (participants affected / at risk) | 75/319 | 129/447 | 140/437
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=319) | Lemborexant 5 mg (N=447) | Lemborexant 10 mg (N=437)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic Retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Jaw Cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Jaw Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic Neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Disturbance In Attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hydrosalpinx (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Floppy eyelid syndrome (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intentional Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (7) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=319) | Lemborexant 5 mg (N=447) | Lemborexant 10 mg (N=437)
Influenza (Infections and infestations) | 15 (15) | 22 (22) | 26 (29)
Nasopharyngitis (Infections and infestations) | 40 (43) | 51 (67) | 48 (56)
Headache (Nervous system disorders) | 21 (33) | 43 (76) | 32 (41)
Somnolence (Nervous system disorders) | 5 (5) | 38 (44) | 60 (64)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT02952820/Prot_002.pdf
  • Statistical Analysis Plan (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT02952820/SAP_003.pdf